CLINICAL TRIAL: NCT01125020
Title: Impact of Postoperative Adjuvant Chemotherapy in Patients With Hepatocellular Carcinoma After Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Changzheng Hospital (Other)
Responsible Party: Shanghai First People's Hosptial
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008BAI60B03
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Last update posted 2010-05-18 (Estimated); Status verified 2010-05

CONDITIONS: Liver Transplantation; Hepatocellular Carcinoma; Tumor Recurrence and Metastasis; Survival; Adjuvant Chemotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence; Neoplasm Metastasis | interventions — Gemcitabine; Oxaliplatin; Doxorubicin; Fluorouracil; Cisplatin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- gemcitabine and oxaliplatin (Active Comparator)
  Interventions: Drug: gemcitabine and oxaliplatin
- doxorubicin, 5-Fu and cisplatin (Active Comparator)
  Interventions: Drug: doxorubicin, 5-Fu and cisplatin

INTERVENTIONS:
Drug: gemcitabine and oxaliplatin — Gemcitabine 1000mg/m2 (days l, 8) and oxaliplatin 130mg/m2 (day l) delivered as an intravenous infusion, given every 28days and repeat six times.
  Arms: gemcitabine and oxaliplatin
Drug: doxorubicin, 5-Fu and cisplatin — Doxorubicin 20mg/m2 (days 1, 3), 5-Fu 300mg/m2 (days 1-5) and cisplatin 20mg/m2 (days 1-3) delivered as an intravenous infusion, given every 28days and repeat six times.
  Arms: doxorubicin, 5-Fu and cisplatin

SUMMARY:
The study is designed to investigate the effect of postoperative adjuvant chemotherapy in prevention of tumor recurrence and metastasis for hepatocellular carcinoma after liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* All liver transplantation patients with hepatocellular carcinoma between Dec 2008 and May 2010 are potentially eligible for enrollment.

Exclusion Criteria:

* Age less than 18 years
* Treatment with other postoperative adjuvant chemotherapy
* Survival is less than 3 months after liver transplantation
* Inability to provide written informed consent prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-05 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
tumor recurrence and metastasis | within the first year after liver transplantation
  Examination of tumor recurrence include serum levels of alpha-fetoprotein(AFP), chest radiography, abdominal ultrasonography, chest or abdominal computed tomography (CT), magnetic resonance imaging (MRI) and bone scintigraphy

SECONDARY OUTCOMES:
Postoperative survival | within the first year after liver transplantation
  Postoperative survival include rates of disease-free survival (DFS), overall survival(OS), tumor recurrence and death.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Hai Peng, MD, Study Chair — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai First People's Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Dudek K, Kornasiewicz O, Remiszewski P, Kobryn K, Ziarkiewicz-Wroblewska B, Gornicka B, Zieniewicz K, Krawczyk M. Impact of tumor characteristic on the outcome of liver transplantation in patients with hepatocellular carcinoma. Transplant Proc. 2009 Oct;41(8):3135-7. doi: 10.1016/j.transproceed.2009.08.016. PMID 19857695
- [Background] Soderdahl G, Backman L, Isoniemi H, Cahlin C, Hockerstedt K, Broome U, Makisalo H, Friman S, Ericzon BG. A prospective, randomized, multi-centre trial of systemic adjuvant chemotherapy versus no additional treatment in liver transplantation for hepatocellular carcinoma. Transpl Int. 2006 Apr;19(4):288-94. doi: 10.1111/j.1432-2277.2006.00279.x. PMID 16573544
- [Background] Louafi S, Boige V, Ducreux M, Bonyhay L, Mansourbakht T, de Baere T, Asnacios A, Hannoun L, Poynard T, Taieb J. Gemcitabine plus oxaliplatin (GEMOX) in patients with advanced hepatocellular carcinoma (HCC): results of a phase II study. Cancer. 2007 Apr 1;109(7):1384-90. doi: 10.1002/cncr.22532. PMID 17330837